CLINICAL TRIAL: NCT01144104
Title: Targeted and Tailored Messages to Enhance Depression Care
Brief Title: Activating Messages for Enhancing Primary Care Practice (AMEP2): Effectiveness Study
Acronym: AMEP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 200917591; 1R01MH079387-01A1 (NIH)
Record Dates: First submitted 2010-05-14; First posted 2010-06-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Public Service Announcements (Experimental): Demographically targeted public service announcement
  Interventions: Behavioral: Public Service Announcement
- Interactive Multi-Media Computer Program (Experimental): Personally tailored information about seeking care for depression based on respondent characteristics
  Interventions: Behavioral: Interactive Multi-Media Computer Program
- Attention Control Video (Active Comparator): Two-minute video focusing on common sleep disorders.
  Interventions: Behavioral: Sleep Hygiene Video

INTERVENTIONS:
Behavioral: Public Service Announcement
  Arms: Public Service Announcements
Behavioral: Interactive Multi-Media Computer Program
  Arms: Interactive Multi-Media Computer Program
Behavioral: Sleep Hygiene Video
  Arms: Attention Control Video

SUMMARY:
This trial consists of two linked substudies.

Substudy 1: Activating Messages for Enhancing Primary Care Practice (AMEP2): Effectiveness Study

Substudy 2: Activating Messages for Enhancing Primary Care Practice (AMEP2): Toxicity Study

The purpose of the Effectiveness Study is to assess the comparative effectiveness of three multimedia educational interventions (a targeted educational video, a tailored interactive multimedia computer program, and an "attention control") for increasing the likelihood that primary care patients with significant depressive symptoms will seek appropriate care (n = 510). The primary study outcomes are provision of minimally acceptable initial care, reductions in depression-related stigma, and improvement in depression symptoms. (See Process of Care and Patient Outcomes in Primary Outcome Measure section.)

The purpose of the Toxicity Study is to assess the potential benefits (reduced stigma) and harms (inappropriate prescribing) associated with three multimedia depression educational interventions when administered to patients with few or no depressive symptoms (n = 308). The primary outcomes relating to this outcome are reducing depression-related stigma and reducing unnecessary prescribing. (See Toxicity in Primary Outcome Measure section.)

Both studies will look at the secondary outcome measure of patient requests for depression treatment.

DETAILED DESCRIPTION:
This project is an investigator-initiated study involving two sequential phases and is funded by the National Institute of Mental Health. Phase I included the use of marketing research (i.e. focus groups, adaptive conjoint analysis, and other survey methods) to produce two clinic-based interventions: a public service announcement (PSA) and interactive multimedia computer program (IMCP). The two clinic-based interventions are intended to include messages that will activate patients to talk with their physicians about specific health concerns (depression) and/or any depressive symptoms they've been experiencing. In Phase II (as described in this registration protocol), those interventions will undergo assessment in a randomized controlled effectiveness trial (RCT) in primary care settings in Sacramento and San Francisco.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70
* Visual acuity and manual dexterity to operate a laptop computer

Exclusion Criteria:

* Currently being treated for depression with anti-depressant medications

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 925 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Process of Care | Within 24 hours of intervention delivery (physician post-visit assessment)
  Minimally acceptable initial care, meaning 1) antidepressant prescription, 2) referral to a mental health specialist, or 3) follow up within 14 days if PHQ >= 15 or within 30 days otherwise
Patient Outcomes | Stigma: Within 24 hours of intervention delivery (patient post-visit assessment); depression symptoms: 12 weeks
  1) Stigma as measured by a scale adapted from Kanter JW, Rusch LC, Brondino MJ. Depression self-stigma: a new measure and preliminary findings. J Nervous Mental Dis 1008; 196(9):663-70, and 2) depression symptoms measured via PHQ-8 scores.
Toxicity | Within 24 hours of intervention delivery (patient and physician post-visit assessment, audio-recording of doctor-patient interaction at index visit)
  1) Stigma as measured by a scale adapted from Kanter (see above) and 2) antidepressant prescribing by physician

SECONDARY OUTCOMES:
Direct or indirect patient requests for depression treatment | Within 24 hours of intervention delivery (physician post-visit assessment, audio-recording of doctor-patient interaction at index visit)
  Patient request for medicine for depression or referral to a mental health professional

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Kravitz, MD, MSPH, Principal Investigator — University of California, Davis; Mitchell L Feldman, MD, MPhil, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - Sutter Health - Elk Grove Family Medicine, Elk Grove, California
  - VA Northern California Healthcare System, Mather, California
  - Kaiser Permanente - Point West, Sacramento, California
  - University of California, Davis, Sacramento, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Derived] Kravitz RL, Franks P, Feldman MD, Tancredi DJ, Slee CA, Epstein RM, Duberstein PR, Bell RA, Jackson-Triche M, Paterniti DA, Cipri C, Iosif AM, Olson S, Kelly-Reif S, Hudnut A, Dvorak S, Turner C, Jerant A. Patient engagement programs for recognition and initial treatment of depression in primary care: a randomized trial. JAMA. 2013 Nov 6;310(17):1818-28. doi: 10.1001/jama.2013.280038. PMID 24193079
- [Derived] Tancredi DJ, Slee CK, Jerant A, Franks P, Nettiksimmons J, Cipri C, Gottfeld D, Huerta J, Feldman MD, Jackson-Triche M, Kelly-Reif S, Hudnut A, Olson S, Shelton J, Kravitz RL. Targeted versus tailored multimedia patient engagement to enhance depression recognition and treatment in primary care: randomized controlled trial protocol for the AMEP2 study. BMC Health Serv Res. 2013 Apr 17;13:141. doi: 10.1186/1472-6963-13-141. PMID 23594572